CLINICAL TRIAL: NCT05179265
Title: A Randomized, Double-blind, Single-dose, Dose-escalated Phase Ia Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of Recombinant Human Serum Albumin in Healthy Subjects
Brief Title: Recombinant Human Serum Albumin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rHSA 2020-1
Record Dates: First submitted 2021-11-02; First posted 2022-01-05 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hepatic Ascites
MeSH Terms: interventions — recombinant human serum albumin-heme; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 0.45 g/bottle，50 mL
  Interventions: Drug: Human serum albumin
- test group (Experimental): 10 g/bottle (20%, 50 mL)
  Interventions: Drug: recombinant human serum albumin

INTERVENTIONS:
Drug: recombinant human serum albumin — 10 g/bottle (20%, 50 mL)
  Arms: test group
Drug: Human serum albumin — 10 g/bottle (20%, 50 mL)
  Arms: Control group

SUMMARY:
This trial adopts a single-center, randomized, double-blind, dose-escalation, placebo-controlled design to evaluate the safety, tolerability, pharmacokinetics, and efficacy of a single administration of recombinant human serum albumin in healthy subjects Kinetics and anti-drug antibody characteristics.

Qualified healthy subjects (both male and female) were screened and enrolled to the four dose levels of 2 g, 5 g, 10 g, and 20 g according to the principle of dose escalation, and 6 out of 8 subjects in each dose group One patient received the test drug, and two received a placebo.

DETAILED DESCRIPTION:
This trial adopts a single-center, randomized, double-blind, dose-escalation, placebo-controlled design to evaluate the safety, tolerability, pharmacokinetics, and efficacy of a single administration of recombinant human serum albumin in healthy subjects Kinetics and anti-drug antibody characteristics.

Qualified healthy subjects (both male and female) were screened and enrolled to the four dose levels of 2 g, 5 g, 10 g, and 20 g according to the principle of dose escalation. 6 out of 8 subjects in each dose group One patient received the test drug, and two received a placebo. Among them, each case in the first dose (2 g) group was enrolled in the group at least 48 hours apart, and was randomly assigned to receive intravenous administration of the test drug or placebo; the first two subjects in the second, third, and fourth dose groups could serve as sentinels. Enrolled at the same time. One patient received the test drug intravenously, the other received a placebo intravenously, and two sentinel subjects completed a single intravenous drug observation for at least 48 hours. If no severe allergic reaction occurred, the group The other subjects in each case were enrolled in the group at least 48 hours apart, and randomly assigned to receive intravenous administration of the test drug or placebo for a single dose of safety, tolerability, pharmacokinetics, and pharmacodynamics And anti-drug antibody test. All subjects should undergo a skin test before receiving the test drug or placebo intravenously, that is, receive an intradermal injection of about 20 mg of the test drug or placebo, and observe the skin test response: if 1 h after the intradermal injection ( ±10 min) If the subject is red, swollen or indurated at the injection site with a diameter of ≤1.5 cm, intravenous administration can be performed, otherwise the subject will have a positive skin test and cannot receive intravenous administration. Subjects who have a positive skin test will withdraw from the test after completing the inspections and operations specified in the protocol. During the test, whether to adjust the positive standard of the skin test reaction will be determined according to the safety information that has been obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 18 to 55 years old (including the critical value), male or female;
2. Body weight ≥45 kg, body mass index (BMI) between 18 and 28 kg/㎡ (including the critical value);
3. Throughout the study period (from screening to 3 months after the end of the study), subjects or their spouses voluntarily use effective contraceptive methods, such as abstinence, condoms, intrauterine device (IUD), and double barrier method (such as condoms and diaphragm), and there was no sperm donation plan for men;
4. Be willing to participate in clinical trials and sign Informed Consent Form;
5. Be able to communicate well with researchers and understand and abide by the requirements of this study.

Exclusion Criteria:

1. Yeast source antibody positive;
2. Investigators consider that there is a clinically significant drug or food allergy, allergic disease history or allergic constitution (≥2 substance allergies), or explicitly allergic to this product or its similar albumin preparation ingredient;
3. History of clinical serious disease, including but not limited to circulatory systems, endocrine systems, gastrointestinal tract, kidneys, nervous systems, blood systems, immune systems, mental disease and metabolic abnormalities, and investigators consider that not suitable for clinical trials ;
4. History of cardiovascular system disease, including but not limited to vital signs abnormalities (such as systolic pressure <90 mmHg or> 140 mmHg, diastolic pressure <50 mmHg or> 90 mmHg, heart rate <50 bpm or> 100 bpm), severe arrhythmia, Heart failure, unstable angina pectoris, myocardial infarction occurred six months prior to screening ､the tachycardia / translucent that needs drug therapy, three-degree atrioventricular block, QTC interval≥450 ms or electrocardiogram has a clinically significant abnormality;
5. Previous has a chronic infectious disease and the investigators can judge possible affecting the evaluation of the drug in trial;
6. Surgery of diseases having clinical significance within 4 weeks before administration;
7. Difficulties with blood collection or cannot be resistant to venipuncture , history of needle sickness or blood sickness.
8. Alcohol breath test , smoke test or drug urinary screening is positive;
9. Physical examination, vital signs, 12 lead electrocardiogram, laboratory examination (blood routine, urine routine, blood biochemical examination, etc.) found that there is a clinical significance;
10. One or more positive results for human immunodeficiency virus (HIV) antibody, treponema pallidum antibody, hepatitis B surface antigen or hepatitis C antibody;
11. A history of drug abuse, or alcohol abuse ( in other words , drinking more than 14 units of alcohol per week [1 unit=360 mL beer or 45 mL of 40% alcoholic spirits or 150 mL wine]) or smoking history (≥5 per day ), or those who cannot smoke during hospitalization;
12. Those who use any caffeine-rich food or beverages (coffee, tea, cola, chocolate, etc.) within 48 hours before the first administration of the study drug, or who do not agree to prohibit the use of caffeine-rich food or beverages during the trial;
13. Those who have special dietary requirements and cannot follow a unified diet;
14. Those who have been treated with corticosteroids or human plasma products within 4 weeks before the trial drug is administered, and have used any prescription drugs, over-the-counter drugs or herbal medicines within 2 weeks (except external preparations or topical preparations);
15. Participated in any drug clinical trial within 3 months before administration;
16. Those who have donated blood within 4 weeks before dosing or plan to donate blood during the study period or within 4 weeks after the end of the study (>400 mL);
17. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial;
18. Researchers believe that compliance is poor, or those who have other factors that are not suitable for participating in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
TEAE | 99 days
  Adverse events will be coded using MedDRA (International Dictionary of Medical Terms)., TEAEs related to test drugs were summarized and analyzed according to SOC and PT, and the number of occurrences and the incidence were calculated.
SAE | 99 days
  Adverse events will be coded using MedDRA (International Dictionary of Medical Terms). SAEs related to test drugs were summarized and analyzed according to SOC and PT, and the number of occurrences and the incidence were calculated.

SECONDARY OUTCOMES:
AUC0-tlast | 57 days
  The PK blood sample collection time point and time window are: within 1 h before intravenous administration, immediately after intravenous administration (+1 min), By collecting within 1 h before intravenous administration, immediately after intravenous administration (+1 min), and after intravenous administration (taking the immediate stop of administration as 0 point) 2 h (± 5 min), 10 h (± 30) min), 24 h (±1 h), 48 h (±1 h), 72 h (±1 h), and D8 (±1 day), D15 (±1 day), D29 (±2 days), D57 (±3 days) blood sample, calculate the PK parameter of the blood sample: AUC0-tlast
Tmax | 57 days
  By collecting within 1 h before intravenous administration, immediately after intravenous administration (+1 min), and after intravenous administration (taking the immediate stop of administration as 0 point) 2 h (± 5 min), 10 h (± 30) min), 24 h (±1 h), 48 h (±1 h), 72 h (±1 h), and D8 (±1 day), D15 (±1 day), D29 (±2 days), D57 (±3 days) blood sample, calculate the PK parameter of the blood sample: Tmax
C0 | 1 day
  The PK blood sample collection time point and time window are: within 1 h before intravenous administration, immediately after intravenous administration (+1 min), and after intravenous administration (take the cessation of administration as the 0 point) 2 h (±5) min), 10 h (±30 min), 24 h (±1 h), 48 h (±1 h), 72 h (±1 h), and D8 (±12 h), D15 (±1 day), D29 (± 2 days), D57 (± 3 days), 2 mL of blood was collected respectively.
C8 | 1 day
  Collect blood samples on the eighth day（±12 h） and determine the albumin concentration on the eighth day
C15 | 1day
  Collect blood samples on the fifteenth day (±1 day)and determine the albumin concentration on the fifteenth day.
C29 | 1 day
  Collect blood samples on the 29th day(±2 days) and determine the albumin concentration on the 29th day.
C57 | 1 day
  Collect blood samples on the 57th day（±3 days） and determine the albumin concentration on the 57th day.
Cmax | 57 days
  By collecting within 1 h before intravenous administration, immediately after intravenous administration (+1 min), and after intravenous administration (taking the immediate stop of administration as 0 point) 2 h (± 5 min), 10 h (± 30) min), 24 h (±1 h), 48 h (±1 h), 72 h (±1 h), and D8 (±1 day), D15 (±1 day), D29 (±2 days), D57 (±3 days) blood sample, calculate the PK parameter of the blood sample: Cmax
Pharmacodynamic analysis | 72 h
  Plasma colloidal osmotic pressure blood sample collection time point: within 1 hour before intravenous administration, immediately after intravenous administration (+1 min), and after intravenous administration (take the immediate stop of administration as the 0 point) 1 hour (±3 min) ), 3 h (± 5 min), 6 h (± 10 min), 24 h (± 1 h), 48 h (± 1 h), 72 h (± 1 h), about 5 hours of blood will be collected at each time point mL.
  Based on the pharmacodynamic analysis set, the statistics of PD indicators of test drugs will be analyzed by descriptive statistical methods.
Evaluate the Anti-Drug antibody (ADA) analysis | 99 days
  The ADA blood sample collection time points are: Day8, Day15, Day29, Day57, and Day99 before the Day1 skin test administration and after the end of the intravenous administration. 6 mL of blood is collected each time, which can be adjusted according to the specific situation. The ADA sample collection time window is the same as the time window of the current visit.
  For subjects who have received the trial drug or placebo intravenously and have at least one valid ADA data, the incidence of rHSA ADA and HCP ADA will be summarized respectively. When ADA is positive, further titer and neutralizing antibody (Nab) analysis can be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bei Hu, Ph.D, Study Director — hubei01_pumch@163.com
Locations (1):
- Shenzheng Protgen Ltd, Guangdong, Shenzheng, China

IPD SHARING:
Plan to Share IPD: No